CLINICAL TRIAL: NCT01121172
Title: Serum Apelin Levels and G212A Polymorphism of Apelin Receptor (APJ)in Obese Children and Adolescents.
Brief Title: Apelin Levels and G212A Polymorphism of Apelin Receptor (APJ)
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Assimina Galli-Tsinopoulou, As. Professor in Pediatric Endocrinology, Aristotle University Of Thessaloniki
Other Study IDs: 10012010
Record Dates: First submitted 2010-05-04; First posted 2010-05-12 (Estimated); Results first posted 2016-05-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-04

CONDITIONS: Obesity; Insulin Resistance; Diabetes Mellitus Type 2
MeSH Terms: conditions — Obesity; Insulin Resistance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- obese: obese subjects according to International Obesity Task Force criteria
- lean

SUMMARY:
The aim of this study is to investigate serum apelin levels as well as their possible association with G212A polymorphism of the apelin receptor in obese children and adolescents.

So far apelin has been reported to be involved in the pathophysiology of various heart diseases such as cardiomyopathies and heart failure. According to recent reports in adults apelin seems to be associated with impaired glucose metabolism, particularly in newly diagnosed diabetes type 2 patients. Obesity is associated with insulin resistance and compensatory hyperinsulinemia leading to diabetes mellitus type 2 even in youngsters. The researchers will try to investigate the role of this new adipokine in order to early detect and to prevent similar entities in childhood obesity.

ELIGIBILITY:
Inclusion Criteria:

* Obese children and adolescents (aged 2-16 years old)

Exclusion Criteria:

* Chronic diseases
* Hypothyroidism
* Medication

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 40 obese children 40 obese adolescents 50 lean children 50 lean adolescents
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2010-05; Primary Completion 2012-06 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Unit of Pediatric Endocrinology, Diabetes and Metabolism-4th Department of Pediatrics, Medical School of Aristotle University of Thessaloniki, Thessaloniki, Greece

RESULTS

PARTICIPANT FLOW:
Groups:
- Obese: obese children and adolescents according to International Obesity Task Force criteria
- Lean: lean children and adolescents matched for age and gender to the obese group
Period: Overall Study
Arm/Group | Obese | Lean
Started | 90 | 90
Completed | 90 | 90
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Obese | Lean | Total
Number analyzed (Participants) | 90 | 90 | 180
Age, Continuous [Median (Full Range); unit: years] | 11.6 [2.6 to 16.5] | 11.7 [3.3 to 17.8] | 11.6 [2.6 to 17.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 47 | 103
  Male | 34 | 43 | 77
Region of Enrollment [Number; unit: participants]
  Greece | 90 | 90 | 180

OUTCOME MEASURES:

1. Primary Outcome: Serum Apelin Levels
Description: Apelin levels were measured in serum of participants, in fasting state
Time Frame: First day after enrollment and after 8-hours of night fasting, at approximately 8:00 pm in the morning
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Obese | Lean
Number analyzed (Participants) | 90 | 90
ng/ml | 1.45 [0.63 to 4.54] | 1.91 [0.55 to 4.71]
Statistical Analysis 1: Comparison: Obese vs Lean; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney); Non parametric test

2. Secondary Outcome: Frequency of G212A Polymorphism of Apelin Receptor in Obese Children and Adolescents
Description: Number of participants with Apelin Receptor Gene G212A polymorphism by genotype group
Time Frame: First day after enrollment
Population: Data were collected only from the Obese participants. Data regarding the genetic polymorphism were not collected from participants forming the Lean Arm/Group.
Measure: Number; unit: participants
Groups:
- Obese Group: Obese children and adolescents according to IOTF criteria
Arm/Group | Obese Group
Number analyzed (Participants) | 90
participants
  GG | 48
  AA | 7
  GA | 35
Statistical Analysis 1: Comparison: Obese Group; Test type: Superiority or Other; p = 0.232, Chi-squared; Chi-square test of frequency distribution amng obese study group and HapMap-CEU polymorphism distribution

ADVERSE EVENTS:
Time Frame: This is a cross-sectional non intervantional, observation study. Time for reporting adverse events was the first day after enrollment, during which blood samples were collected.
Arm/Group | Obese | Lean
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/90
Other Adverse Events (participants affected / at risk) | 0/90 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No